CLINICAL TRIAL: NCT03529864
Title: Effects of Therapeutic Exercise on Health-related Quality of Life and Disability in Students: a Randomized Controlled Trial
Brief Title: Effects of Therapeutic Exercise on Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade da Coruña (Other)
Responsible Party: Principal Investigator, Beatriz Rodríguez-Romero, University Lecturer in the Department of Biomedical Sciences, Medicine and Physiotherapy. University of A Coruña, Universidade da Coruña
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: Experim Fac
Record Dates: First submitted 2018-03-15; First posted 2018-05-18 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Physical Therapy; Health Promotion; Quality of Life
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Why: The design of the intervention took into account the available evidence for the prevention and treatment of neck and low back pain.
  What: Materials: mats, fit-balls, TheraBands, towels, Dyn-Air cushions, chairs, stretchers.
  Procedures: 3 levels of exercises of increasing difficulty. Standing warm-up exercises. Exercises involving: body scanner and breathing pattern re-education (4 minutes), neutral lumbar-pelvic position control in all directions (6 minutes); transverse abdominis activation (4 minutes); neutral cervical position control (2 minutes); global stabilizer activation exercises for the lumbar-pelvic and cervical-scapular regions (4 minutes); low back flexibility (2 minutes); and muscular strengthening and stretching (12 minutes).
  Who provided: Physiotherapist. How: Face to face, group with 8-9 participants.
Masking Description: This study was single-blind, parallel-group, and participants were randomly assigned to either the experimental (EG) or the control group (CG). Randomization was designed after initially evaluating the participants. The EG participated in the progressive exercise therapy program. In contrast, the CG did not receive any type of information or instructions apart from the general information sheet on the progress of the study, attached to the informed consent form.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise therapy (Experimental): The participants took part in a progressive exercise therapy program for 9 consecutive weeks, once a week. This consisted of group sessions with 8 or 9 students, with each session lasting 60 minutes, supervised by the principal researcher
  Interventions: Other: Exercise Therapy
- Control (No Intervention): The CG did not receive any type of information or instructions apart from the general information sheet on the progress of the study, attached to the informed consent form

INTERVENTIONS:
Other: Exercise Therapy
  Arms: Exercise therapy

SUMMARY:
The main objective was to determine the efficacy and safety of a therapeutic exercise program for students. Secondary objectives, determine the prevalence and intensity of musculoskeletal pain (MSP), disability, Health-Related Quality of Life (HRQOL), and satisfaction and perceived improvement with program.

DETAILED DESCRIPTION:
Methodology: randomized, controlled, open clinical trial. Subjects were recruited from students of Degree of Physiotherapy. Inclusion and exclusion criteria were established. Physical Component Summary (PCS) of SF36, as primary outcomes, was taken to the sample size. Randomization was single-blind. Secondary response variables were measured through the Nordic Musculoskeletal Questionnaire, Visual Analogue Scale, Oswestry Disability Index, Neck Disability Index, trunk flexor endurance test and finger-floor distance test. An assessment pre and post intervention was performed. This consisted of a therapeutic exercise program based on the stabilization, 9 sessions of 1 hour. For statistical analysis, the Shapiro-Wilk test, Student's t test or test MannWitney, the statistic (X2) chi-square or Fisher's exact test were applied. The level of significance was taken as p <0.05. Information sheet and informed consent model was delivered.

ELIGIBILITY:
Inclusion Criteria:

* students taking a course of the Physiotherapy Degree
* having enrolled in October 2014
* having given their informed consent.

Exclusion Criteria:

* not accepting to take part in the study,
* not attending the initial evaluation sessions,
* having any type of cardiovascular, neuromusculoskeletal or systemic diseases that restricted exercise participation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-10-03 (Actual); Primary Completion 2014-10-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
SF-36v2 Health Survey | 7 min
  This is self-administered and consists of 36 items that assess the state of health in 8 dimensions: physical function (PF), role-physical (RP), bodily pain (BP), general health (GH), vitality (VT), social function (SF), role-emotional (RE) and mental health (MH). These dimensions may be reduced to 2 scores: Physical Component Summary (PCS) and Mental Component Summary (MCS). In order to interpret the results, standardized scores are obtained with the values for the reference population standards, whereby a score of 50 (SD = 10) represented the mean for the general population, and a score of 10 was one standard deviation. Values over or below 50 have to be respectively interpreted as better or worse than those of the reference population.

SECONDARY OUTCOMES:
Nordic Musculoskeletal Questionnaire (NMQ-E) | 4 min
  It collects information regarding the onset, prevalence, and consequences of musculoskeletal pain. It inquires about ''ache, pain or discomfort'' and 9 body regions are visually depicted on a body chart. In total, it is comprised of 11 questions, equating to 99 data items generated by the tool. With the exception of age data, all response options are dichotomous (yes/no). Questions are ordered in such a way that those relating to the respondents' lifetime (''ever'') are asked first, followed by prevalence questions, and lastly items relating to consequences of pain in the previous year. Respondents are asked to answer all questions for a body region before progressing to the next region (horizontally). In 2 instances (specifically, questions relating to lifetime and annual prevalence of trouble), if the respondent answer no, they are directed to go on to the next body region and all remaining questions for that region are automatically coded as negative responses.
Visual Analogy Scale (VAS) | 2 min
  The pain VAS is a single-item scale. It is a continuous scale comprised of a horizontal line, 10 centimetres (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme: "no pain" (score of 0) and "worst imaginable pain" (score of 100 [100-mm scale]). Although there are no normative values, the recommended cut-off points were used to interpret the score obtained on this scale: no pain (0-4 mm), slight pain (5-44 mm), moderate pain (45-74 mm) and severe pain (75-100 mm) (Hawker GA et al. 2011).
Oswestry Disability Index (ODI) | 4 min
  Lumbar disability
Neck Disability Index (NDI) | 4 min
  Neck disability
Flexor trunk endurance test | 10 min
  Abdominal muscle endurance

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoy D, March L, Brooks P, Blyth F, Woolf A, Bain C, Williams G, Smith E, Vos T, Barendregt J, Murray C, Burstein R, Buchbinder R. The global burden of low back pain: estimates from the Global Burden of Disease 2010 study. Ann Rheum Dis. 2014 Jun;73(6):968-74. doi: 10.1136/annrheumdis-2013-204428. Epub 2014 Mar 24. PMID 24665116
- [Background] Hoy D, March L, Woolf A, Blyth F, Brooks P, Smith E, Vos T, Barendregt J, Blore J, Murray C, Burstein R, Buchbinder R. The global burden of neck pain: estimates from the global burden of disease 2010 study. Ann Rheum Dis. 2014 Jul;73(7):1309-15. doi: 10.1136/annrheumdis-2013-204431. Epub 2014 Jan 30. PMID 24482302
- [Background] Steffens D, Maher CG, Pereira LS, Stevens ML, Oliveira VC, Chapple M, Teixeira-Salmela LF, Hancock MJ. Prevention of Low Back Pain: A Systematic Review and Meta-analysis. JAMA Intern Med. 2016 Feb;176(2):199-208. doi: 10.1001/jamainternmed.2015.7431. PMID 26752509
- [Background] Gross AR, Paquin JP, Dupont G, Blanchette S, Lalonde P, Cristie T, Graham N, Kay TM, Burnie SJ, Gelley G, Goldsmith CH, Forget M, Santaguida PL, Yee AJ, Radisic GG, Hoving JL, Bronfort G; Cervical Overview Group. Exercises for mechanical neck disorders: A Cochrane review update. Man Ther. 2016 Aug;24:25-45. doi: 10.1016/j.math.2016.04.005. Epub 2016 Apr 20. PMID 27317503